CLINICAL TRIAL: NCT03766113
Title: Effect of Unimodal (EEG) and Bimodal (EEG-fMRI) Neurofeedback on Upper Limb Recovery After Stroke
Brief Title: Neurofeedback for Upper-limb Recovery After Stroke
Acronym: NeuroFB-AVC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 35RC18_9813_NeuroFB-AVC
Record Dates: First submitted 2018-11-22; First posted 2018-12-06 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: Neurofeedback ; fMRI ; EEG ; BCI ; Motor imagery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteer (Other): * 50 subjects
  * A single neurofeedback coupling electroencephalogram and functional MRI in time actual .
  Interventions: Other: Neurofeedback coupling electroencephalogram and functional MRI in time actual
- Patients at the early stage after stroke (Other): * 30 subjects
  * Effectiveness of an electroencephalogram-neurofeedback
  Interventions: Other: Electroencephalogram-neurofeedback program or Neurofeedback-free mental imaging program with electroencephalogram recording
- Patients at the chronic stage after stroke (Other): * 36 subjects
  * Effectiveness of a neurofeedback coupling electroencephalogram and functional MRI in time actual
  Interventions: Other: Neurofeedback coupling electroencephalogram and functional MRI in time actual or a neurofeedback-free mental imaging program with electroencephalogram recording

INTERVENTIONS:
Other: Neurofeedback coupling electroencephalogram and functional MRI in time actual — One visit : Neurofeedback coupling electroencephalogram and functional MRI in time actual
  Arms: Healthy volunteer
Other: Electroencephalogram-neurofeedback program or Neurofeedback-free mental imaging program with electroencephalogram recording — Interventional group (Electroencephalogram-neurofeedback program) : 24 minutes, 3 times a week for 12 weeks in addition to the traditional rehabilitation program.
  Controle Group (Neurofeedback-free mental imaging) : 24 minutes, 3 times a week for 12 weeks in addition to the traditional rehabilitation program of reference.
  Arms: Patients at the early stage after stroke
Other: Neurofeedback coupling electroencephalogram and functional MRI in time actual or a neurofeedback-free mental imaging program with electroencephalogram recording — Interventional group (5 weeks) : 5 sessions of neurofeedback coupling electroencephalogram and functional MRI in time actual and 9 sessions of electroencephalogram-neurofeedback program
  Controle Group (5 weeks) : 14 sessions of neurofeedback-free mental imaging program
  Arms: Patients at the chronic stage after stroke

SUMMARY:
Interventional study with minimal risks and constraints, prospective, monocentric.

DETAILED DESCRIPTION:
Neurofeedback (NF) consists on training self-regulation of brain activity by providing real-time information about the participant brain function NF approaches in stroke are usually based on real-time monitoring of brain activity using EEG-NF and involve chronic stroke. Recent studies have revealed the potential of combining EEG and fMRI to achieve a more efficient and specific self-regulation, which may be critical in clinical applications.

The aim of this study is to optimize the neurofeedback method coupling EEG and fMRI in healthy subjects then to evaluate the effect of an EEG-NF and a neurofeedback coupling EEG and fMRI versus motor imagery on recovery in the early and chronic stage after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the early stage after stroke : Ischemic or hemorrhagic unilateral stroke ; adult (age greater than or equal to 18 years) under 80, of both sexes ; stroke less than 1 month old ; upper limb deficit defined by a SAFE score <8 (SAFE Stinear protocol) at D3 of stroke; absence of comprehension difficulties limiting participation ; with or without homonymous lateral hemianopia ; with or without visuospatial henegligence ; free, informed and written consent signed by the patient or a member of his entourage (in the case of a patient able to understand the information and to express his / her consent but presenting motor difficulties leading to an invalid signature).
* Patients at the chronic stage after stroke : Ischemic or unilateral supra-tentorial unilateral cerebral hemorrhage ; adult (age greater than or equal to 18 years) under 80, of both sexes ; stroke more than 6 months ; motor abilities of the upper limb defines as "poor" to "noticeable" according to Hoonhorst on the Fugl-Meyer upper limb scale, ranging between 22 and 53 out of 66 ; absence of comprehension difficulties limiting participation ; with or without homonymous lateral hemianopia ; with or without visuospatial henegligence ; free, informed and written consent signed by the patient or a member of his entourage (in the case of a patient able to understand the information and to express his / her consent but presenting motor difficulties leading to an invalid signature).
* Healthy Volunteers : Adult (age greater than or equal to 18 years) under 80, of both sexes ; Free, informed and written consent signed by the volunteer.

Exclusion Criteria:

* Patients at the early stage after stroke : Ischemic or haemorrhagic involvement of the brainstem ; multiple stroke ; aphasia with major comprehension disorder ; major persons subject to legal protection, persons deprived of their liberty.
* Patients at the chronic stage after stroke : Ischemic or haemorrhagic involvement of the brainstem ; multiple stroke ; aphasia with major comprehension disorder ; vascular leukopathy important to MRI (Fazekas 3) in order not to interfere with the interpretation of MRI ; contraindication to MRI ; major persons subject to legal protection, persons deprived of their liberty.
* Healthy Volunteers : Contraindication to MRI ; pregnancy ; breastfeeding ; major persons subject to legal protection, persons deprived of their liberty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
CXa: Active range of motion at elbow and wirst (from Tardieu scale) | Change in Cxa between baseline and the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Simon Butet, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France